CLINICAL TRIAL: NCT00196794
Title: A Randomized, Double-Blind Study of GT267-004 Versus Vancomycin, and GT267-004 Versus Metronidazole in Patients With C. Difficile-Associated Diarrhea
Brief Title: A Study of GT267-004 Versus Vancomycin and GT267-004 Versus Metronidazole in Patients With C. Difficile-Associated Diarrhea
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Genzyme, a Sanofi Company (Industry)
Responsible Party: Medical Monitor, Genzyme Corporation
Organization: Sanofi (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GD3-170-302
Record Dates: First submitted 2005-09-13; First posted 2005-09-20 (Estimated); Last update posted 2014-03-19 (Estimated); Status verified 2014-03

CONDITIONS: Clostridium Enterocolitis; Diarrhea
Keywords: Pseudomembranous Colitis; Clostridium difficile-associated diarrhea; C. difficile; CDAD
MeSH Terms: conditions — Enterocolitis, Pseudomembranous; Diarrhea

INTERVENTIONS:
Drug: Tolevamer potassium-sodium (GT267-004)

SUMMARY:
Approximately 520 patients will be entered into this study taking place throughout Australia and Europe. This study aims to determine if an investigational drug is safe and effective for treating symptoms of C. difficile-associated diarrhea (CDAD) and lowering the risk of repeat episodes of CDAD. The investigational drug will be evaluated in comparison to current standard antibiotic treatment, so all patients will receive active medication. All study related care is provided including doctor visits, physical exams, laboratory tests, and study medication. The total length of participation is approximately 6 weeks.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age and above
* The presence of CDAD at the time of enrollment with no other likely etiology for the diarrhea
* Less than or equal to 48 hours of treatment with metronidazole, vancomycin or other antibacterial therapy specific for CDAD
* Baseline serum potassium > 3.0 mmol (meq)/L
* Patient considered sufficiently stable clinically to likely complete 6 week study period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 520 (Actual)
Dates: Start 2005-04; Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
Resolution of diarrhea

SECONDARY OUTCOMES:
Time to resolution of diarrhea
Recurrence rate
Number of stools
Average stool consistency
Treatment success

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Genzyme, a Sanofi Company
Locations (118):
- Australia (18):
  - Adelaide
  - Bedford Park
  - Cairns
  - Concord
  - Darlinghurst
  - Five Dock
  - Footscray
  - Herston
  - Hobart
  - Kogarah
  - Nambour
  - Nedlands
  - Parkville
  - Perth
  - Randwick
  - South Brisbane
  - Southport
  - Woolloongabba
- Austria (4):
  - Innsbruck
  - Linz
  - Oberndorf
  - Salzburg
- Belgium (7):
  - Aalst
  - Braine-l'Alleud
  - Brussels
  - Ghent
  - Hasselt
  - Leuven
  - Yvoir
- Czechia (5):
  - Brno
  - Hradec Králové
  - Mělník
  - Ostrava
  - Prague
- Denmark (3):
  - Copenhagen
  - Herlev
  - Hvidovre
- France (11):
  - Amiens
  - Annecy
  - Clichy
  - Créteil
  - Dijon
  - Garches
  - Nice
  - Paris
  - Saint-Etienne
  - Tourcoing
  - Vandœuvre-lès-Nancy
- Germany (12):
  - Augsburg
  - Berlin
  - Cologne
  - Düsseldorf
  - Frankfurt
  - Greifswald
  - Hanover
  - Hofheim
  - Leipzig
  - Lübeck
  - Regensburg
  - Wilhelmshaven
- Ireland (3):
  - Castlebar
  - Cork
  - Dublin
- Norway (7):
  - Bergen
  - Bodø
  - Oslo
  - Stavanger
  - Tromsø
  - Trondheim
  - Tønsberg
- Portugal (4):
  - Carnaxide
  - Coimbra
  - Matosinhos Municipality
  - Porto
- Spain (13):
  - Alcalá de Henares
  - Badalona
  - Barcelona
  - Córdoba
  - Donostia / San Sebastian
  - El Palmar-Murcia
  - Guadalajara
  - Leganés
  - Lleida
  - Madrid
  - Santander
  - Seville
  - Terrassa
- Sweden (9):
  - Gothenburg
  - Jönköping
  - Kalmar
  - Karlskrona
  - Kristianstad
  - Lund
  - Malmo
  - Örebro
  - Skövde
- Switzerland (5):
  - Baden
  - Basel
  - Bellinzona
  - Geneva
  - Lugano
- United Kingdom (17):
  - Abergavenny
  - Birmingham
  - Bristol
  - Bury
  - Cardiff
  - Edinburgh
  - Gwent
  - Ipswich
  - Keighley
  - Leeds
  - Liverpool
  - London
  - Salford
  - Sheffield
  - Stockport
  - Sunderland
  - Winchester

REFERENCES:
- [Derived] Johnson S, Louie TJ, Gerding DN, Cornely OA, Chasan-Taber S, Fitts D, Gelone SP, Broom C, Davidson DM; Polymer Alternative for CDI Treatment (PACT) investigators. Vancomycin, metronidazole, or tolevamer for Clostridium difficile infection: results from two multinational, randomized, controlled trials. Clin Infect Dis. 2014 Aug 1;59(3):345-54. doi: 10.1093/cid/ciu313. Epub 2014 May 5. PMID 24799326